CLINICAL TRIAL: NCT03065530
Title: Efficacy and Safety of Dexmedetomidine Combined With Butorphanol Tartrate for Postoperative Analgesia and Breastfeeding in Cesarean Section
Brief Title: Intravenous Dexmedetomidine for Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shijiang Liu, Attending, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-SR-203
Record Dates: First submitted 2017-02-18; First posted 2017-02-28 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Breast Feeding; Analgesia Obstetrical; Postoperative Pain
Keywords: Dexmedetomidine; Butorphanol tartrate; Analgesia; Breastfeeding; Relative infant dose
MeSH Terms: conditions — Breast Feeding; Pain, Postoperative; Agnosia | interventions — Saline Solution; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Placebo Comparator): The placebo group will pumped in the same volume of saline 0.9% as calculated by parturients' weight in 30 min and receive 1mg butorphanol after delivery.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Interventions: Drug: Normal Saline
- Dexmedetomidine 0.03ug/kg/h group (Experimental): This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min and 1mg butorphanol tartrate after delivery.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.03ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Interventions: Drug: Dexmedetomidine 0.03ug/kg/h
- Dexmedetomidine 0.05ug/kg/h group (Experimental): This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min and 1mg butorphanol tartrate after delivery.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.05ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Interventions: Drug: Dexmedetomidine 0.05ug/kg/h
- Dexmedetomidine 0.08ug/kg/h group (Experimental): This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min and 1mg butorphanol tartrate after delivery.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.08ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Interventions: Drug: Dexmedetomidine 0.08ug/kg/h

INTERVENTIONS:
Drug: Normal Saline — Drug: Normal saline control group receive NS after delivery. Drug: butorphanol tartrate PCA: butorphanol tartrate after cesarean section.
  Arms: control group
Drug: Dexmedetomidine 0.03ug/kg/h — Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.03ug/kg/h Dexmedetomidine after cesarean section.
  Other Names: dexmedetomidine Injection; Dexmedetomidine Hydrochloride
  Arms: Dexmedetomidine 0.03ug/kg/h group
Drug: Dexmedetomidine 0.05ug/kg/h — Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.05ug/kg/h Dexmedetomidine after cesarean section.
  Other Names: dexmedetomidine Injection; Dexmedetomidine Hydrochloride
  Arms: Dexmedetomidine 0.05ug/kg/h group
Drug: Dexmedetomidine 0.08ug/kg/h — Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.08ug/kg/h Dexmedetomidine after cesarean section.
  Other Names: dexmedetomidine Injection; Dexmedetomidine Hydrochloride
  Arms: Dexmedetomidine 0.08ug/kg/h group

SUMMARY:
Nervous, anxiety, fear and other psychological reactions always appears in parturients during cesarean section. This study intends to investigate the effectiveness and safety of dexmedetomidine combined with butorphanol tartrate for postoperative analgesia and breastfeeding after caesarean section.

ELIGIBILITY:
Inclusion Criteria:

1. Parturients who had successfully breastfed a prior infant and planned to breastfeed after this delivery were screened for eligibility.
2. Parturients undergoing elective caesarean delivery under epidural anaesthesia
3. ASA I and II parturients aged 18-45 years, with singleton gestation.
4. Parturients with verbal and written mandarin
5. Parturients who want to use PCA intravenous analgesia and can use the pump correctly
6. written informed consent.

Exclusion Criteria

1. Multiple gestation.
2. A history of allergy to dexmedetomidine or other study drugs
3. Cardiovascular disease (basic HR<50bpm or SBP<100mmHg)
4. Opioid drugs abuse.
5. BMI more than 35 kg/m2
6. Conditions that preclude spinal anesthesia.
7. Preeclampsia or epilepsy.
8. A history of neuromuscular disease.
9. Epidural anaesthesia was unsuccessful.
10. The parturients, whose surgery ended after 11 a.m.

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Result] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Result] Kainu JP, Halmesmaki E, Korttila KT, Sarvela PJ. Persistent Pain After Cesarean Delivery and Vaginal Delivery: A Prospective Cohort Study. Anesth Analg. 2016 Dec;123(6):1535-1545. doi: 10.1213/ANE.0000000000001619. PMID 27870738
- [Result] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Result] Lin TF, Yeh YC, Lin FS, Wang YP, Lin CJ, Sun WZ, Fan SZ. Effect of combining dexmedetomidine and morphine for intravenous patient-controlled analgesia. Br J Anaesth. 2009 Jan;102(1):117-22. doi: 10.1093/bja/aen320. Epub 2008 Nov 5. PMID 18987053
- [Result] Jakob SM, Ruokonen E, Grounds RM, Sarapohja T, Garratt C, Pocock SJ, Bratty JR, Takala J; Dexmedetomidine for Long-Term Sedation Investigators. Dexmedetomidine vs midazolam or propofol for sedation during prolonged mechanical ventilation: two randomized controlled trials. JAMA. 2012 Mar 21;307(11):1151-60. doi: 10.1001/jama.2012.304. PMID 22436955
- [Result] Schnabel A, Meyer-Friessem CH, Reichl SU, Zahn PK, Pogatzki-Zahn EM. Is intraoperative dexmedetomidine a new option for postoperative pain treatment? A meta-analysis of randomized controlled trials. Pain. 2013 Jul;154(7):1140-9. doi: 10.1016/j.pain.2013.03.029. Epub 2013 Mar 27. PMID 23706726
- [Result] Colin PJ, Hannivoort LN, Eleveld DJ, Reyntjens KMEM, Absalom AR, Vereecke HEM, Struys MMRF. Dexmedetomidine pharmacokinetic-pharmacodynamic modelling in healthy volunteers: 1. Influence of arousal on bispectral index and sedation. Br J Anaesth. 2017 Aug 1;119(2):200-210. doi: 10.1093/bja/aex085. PMID 28854538
- [Result] Arain SR, Ruehlow RM, Uhrich TD, Ebert TJ. The efficacy of dexmedetomidine versus morphine for postoperative analgesia after major inpatient surgery. Anesth Analg. 2004 Jan;98(1):153-158. doi: 10.1213/01.ANE.0000093225.39866.75. PMID 14693611
- [Result] Ren C, Chi M, Zhang Y, Zhang Z, Qi F, Liu Z. Dexmedetomidine in Postoperative Analgesia in Patients Undergoing Hysterectomy: A CONSORT-Prospective, Randomized, Controlled Trial. Medicine (Baltimore). 2015 Aug;94(32):e1348. doi: 10.1097/MD.0000000000001348. PMID 26266386
- [Result] Orbach-Zinger S, Fireman S, Ben-Haroush A, Karoush T, Klein Z, Mazarib N, Artyukh A, Chen R, Ioscovich A, Eidelman LA, Landau R. Preoperative sleep quality predicts postoperative pain after planned caesarean delivery. Eur J Pain. 2017 May;21(5):787-794. doi: 10.1002/ejp.980. Epub 2016 Dec 15. PMID 27977073
- [Result] Hsu YW, Cortinez LI, Robertson KM, Keifer JC, Sum-Ping ST, Moretti EW, Young CC, Wright DR, Macleod DB, Somma J. Dexmedetomidine pharmacodynamics: part I: crossover comparison of the respiratory effects of dexmedetomidine and remifentanil in healthy volunteers. Anesthesiology. 2004 Nov;101(5):1066-76. doi: 10.1097/00000542-200411000-00005. PMID 15505441
- [Result] El-Tahan MR, Mowafi HA, Al Sheikh IH, Khidr AM, Al-Juhaiman RA. Efficacy of dexmedetomidine in suppressing cardiovascular and hormonal responses to general anaesthesia for caesarean delivery: a dose-response study. Int J Obstet Anesth. 2012 Jul;21(3):222-9. doi: 10.1016/j.ijoa.2012.04.006. Epub 2012 Jun 7. PMID 22681971
- [Result] Nie Y, Liu Y, Luo Q, Huang S. Effect of dexmedetomidine combined with sufentanil for post-caesarean section intravenous analgesia: a randomised, placebo-controlled study. Eur J Anaesthesiol. 2014 Apr;31(4):197-203. doi: 10.1097/EJA.0000000000000011. PMID 24463478
- [Result] Sia AT, Sng BL. Intravenous dexmedetomidine for obstetric anaesthesia and analgesia: converting a challenge into an opportunity? Int J Obstet Anesth. 2009 Jul;18(3):204-6. doi: 10.1016/j.ijoa.2009.02.008. Epub 2009 May 22. No abstract available. PMID 19464877
- [Result] Abu-Halaweh SA, Al Oweidi AK, Abu-Malooh H, Zabalawi M, Alkazaleh F, Abu-Ali H, Ramsay MA. Intravenous dexmedetomidine infusion for labour analgesia in patient with preeclampsia. Eur J Anaesthesiol. 2009 Jan;26(1):86-7. doi: 10.1097/EJA.0b000e000000f3fb. No abstract available. PMID 19122562
- [Result] Nakanishi R, Yoshimura M, Suno M, Yamamoto K, Ito H, Uchimine Y, Toriumi T, Kurosawa A, Sugawara A, Kunisawa T. Detection of dexmedetomidine in human breast milk using liquid chromatography-tandem mass spectrometry: Application to a study of drug safety in breastfeeding after Cesarean section. J Chromatogr B Analyt Technol Biomed Life Sci. 2017 Jan 1;1040:208-213. doi: 10.1016/j.jchromb.2016.11.015. Epub 2016 Nov 10. PMID 27856195
- [Result] Yoshimura M, Kunisawa T, Suno M, Sugawara A, Kurosawa A, Nakanishi R, Aoki K, Toriumi T. Intravenous dexmedetomidine for cesarean delivery and its concentration in colostrum. Int J Obstet Anesth. 2017 Nov;32:28-32. doi: 10.1016/j.ijoa.2017.05.002. Epub 2017 May 10. PMID 28687146
- [Result] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Result] Wang C, Liu S, Han C, Yu M, Hu Y, Liu C. Effect and placental transfer of dexmedetomidine during caesarean section under epidural anaesthesia. J Int Med Res. 2017 Jun;45(3):964-972. doi: 10.1177/0300060517698330. Epub 2017 Apr 28. PMID 28449631
- [Result] Jiang W, Wang Q, Xu M, Li Y, Yang R, Song X, Duan H, Zhang P. Assessment of different loading doses of dexmedetomidine hydrochloride in preventing adverse reaction after combined spinal-epidural anesthesia. Exp Ther Med. 2017 Jun;13(6):2946-2950. doi: 10.3892/etm.2017.4335. Epub 2017 Apr 13. PMID 28587365
- [Result] Chen Z, Tang R, Zhang R, Jiang Y, Liu Y. Effects of dexmedetomidine administered for postoperative analgesia on sleep quality in patients undergoing abdominal hysterectomy. J Clin Anesth. 2017 Feb;36:118-122. doi: 10.1016/j.jclinane.2016.10.022. Epub 2016 Dec 1. PMID 28183547
- [Result] Deussen AR, Ashwood P, Martis R. Analgesia for relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2011 May 11;(5):CD004908. doi: 10.1002/14651858.CD004908.pub2. PMID 21563142
- [Result] Kelly LE, Chaudhry SA, Rieder MJ, 't Jong G, Moretti ME, Lausman A, Ross C, Berger H, Carleton B, Hayden MR, Madadi P, Koren G. A clinical tool for reducing central nervous system depression among neonates exposed to codeine through breast milk. PLoS One. 2013 Jul 29;8(7):e70073. doi: 10.1371/journal.pone.0070073. Print 2013. PMID 23922910
- [Result] Chow CK, Koren G. Sedating drugs and breastfeeding. Can Fam Physician. 2015 Mar;61(3):241-3. PMID 25927109
- [Result] Newton ER, Hale TW. Drugs in Breast Milk. Clin Obstet Gynecol. 2015 Dec;58(4):868-84. doi: 10.1097/GRF.0000000000000142. PMID 26457856
- [Result] Anttila M, Penttila J, Helminen A, Vuorilehto L, Scheinin H. Bioavailability of dexmedetomidine after extravascular doses in healthy subjects. Br J Clin Pharmacol. 2003 Dec;56(6):691-3. doi: 10.1046/j.1365-2125.2003.01944.x. PMID 14616431
- [Result] Lind JN, Perrine CG, Li R. Relationship between use of labor pain medications and delayed onset of lactation. J Hum Lact. 2014 May;30(2):167-73. doi: 10.1177/0890334413520189. Epub 2014 Jan 22. PMID 24451212
- [Result] Sia AT, Kwek K, Yeo GS. The in vitro effects of clonidine and dexmedetomidine on human myometrium. Int J Obstet Anesth. 2005 Apr;14(2):104-7. doi: 10.1016/j.ijoa.2004.11.004. PMID 15795144
- [Result] Yu M, Han C, Jiang X, Wu X, Yu L, Ding Z. Effect and Placental Transfer of Dexmedetomidine During Caesarean Section Under General Anaesthesia. Basic Clin Pharmacol Toxicol. 2015 Sep;117(3):204-8. doi: 10.1111/bcpt.12389. Epub 2015 Mar 4. PMID 25652672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parturients (>18 and <45 years old) with a singleton pregnancy admitted to our institute who underwent elective caesarean delivery under epidural anaesthesia were recruited in this study between February 2017 and October 2017.
Pre-assignment Details: not meeting inclusion criteria (n=39)
  declined to participate , n=14
  other reasons, n=3
Groups:
- Group C: The placebo group will pumped in the same volume of saline 0.9% as calculated by parturients' weight in 30 min.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Normal Saline: Drug: Normal saline control group receive NS after delivery. Drug: butorphanol tartrate PCA: butorphanol tartrate after cesarean section.
- Group D1: This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.03ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Dexmedetomidine 0.03ug/kg/h: Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.03ug/kg/h Dexmedetomidine after cesarean section.
- Group D2: This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.05ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Dexmedetomidine 0.05ug/kg/h: Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.05ug/kg/h Dexmedetomidine after cesarean section.
- Group D3: This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.08ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Dexmedetomidine 0.08ug/kg/h: Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.08ug/kg/h Dexmedetomidine after cesarean section.
Period: Overall Study
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Started | 30 | 30 | 30 | 30
Completed | 28 | 29 | 29 | 28
Not Completed | 2 | 1 | 1 | 2
Not completed — Lack of Efficacy | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: The placebo group will pumped in the same volume of saline 0.9% as calculated by parturients' weight in 30 min.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Normal Saline: Drug: Normal saline control group receive NS after delivery. Drug: butorphanol tartrate PCA: butorphanol tartrate after cesarean section.
- Dexmedetomidine 0.03ug/kg/h: This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.03ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Dexmedetomidine 0.03ug/kg/h: Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.03ug/kg/h Dexmedetomidine after cesarean section.
- Dexmedetomidine 0.05ug/kg/h: This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.05ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Dexmedetomidine 0.05ug/kg/h: Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.05ug/kg/h Dexmedetomidine after cesarean section.
- Dexmedetomidine 0.08ug/kg/h: This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.08ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Dexmedetomidine 0.08ug/kg/h: Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.08ug/kg/h Dexmedetomidine after cesarean section.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dexmedetomidine 0.03ug/kg/h | Dexmedetomidine 0.05ug/kg/h | Dexmedetomidine 0.08ug/kg/h | Total
Number analyzed (Participants) | 28 | 29 | 29 | 28 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 29 | 28 | 114
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.75 (3.46) | 31.41 (3.69) | 32.07 (4.2) | 31.11 (3.37) | 31.59 (3.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 29 | 28 | 114
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 28 | 29 | 29 | 28 | 114
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 28 | 29 | 29 | 28 | 114

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) at Rest
Description: visual analogue scale (VAS; with 0, no pain; to 10, the worst imaginable pain) is a validated assessing scale for pain intensity. VAS at rest was assessed when the patient was in supine position
Time Frame: 6h after cesarean section.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
units on a scale | 3.143 (1.38) | 2.897 (1.012) | 1.665 (1.045) | 1.25 (0.7515)
Statistical Analysis 1: Comparison: Group C vs Group D1 vs Group D2 vs Group D3; The sample size was calculated on the basis of an our initial pilot study, and the SD was 1.4 between the four groups. We hypothesized that the differences in VAS between the four groups and the SDs would be 15%. A power analysis suggested that there will be 80% power to detect differences at an α=0.05 significance level (two-tailed), including 24 individuals per treatment group. Considering the exclusion of 25% of patients, 30 parturients were eventually recruited in each group; Test type: Other; p < 0.05, Kruskal-Wallis

2. Secondary Outcome: Relative Infant Dose (RID) of Dexmedetomidine
Description: Relative infant dose (RID) =Dose (infant, mg•kg-1•day-1) /Dose (mother, mg•kg-1•day-1) μg·kg-1·h-1. The Dose (infant) in mg•kg-1 is calculated by multiplying the concentration of the drug in breast milk by the volume of breast milk consumed daily (about 150 mL•kg-1).
Time Frame: 48h after cesarean section.
Measure: Mean (Standard Deviation); unit: percentage of one hundred
Arm/Group | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 16 | 15 | 17
percentage of one hundred | 0.1712 (0.1764) | 0.1967 (0.1141) | 0.3701 (0.2357)

3. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) at Rest
Description: as for outcome 1
Time Frame: 12h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 3.29 (1.01) | 2.86 (0.99) | 1.62 (0.78) | 0.93 (0.94)

4. Secondary Outcome: Ramsay Sedation Score(RSS)
Description: Sedation intensity measured with RSS is recorded at the 6, 12 24 and 48 h after cesarean section. Sedation was assessed by the Ramsay Sedation Scores (RSS) (1, anxious patient; 2, cooperative and tranquil; 3, responding to command; 4, brisk response to stimulus; 5, sluggish response to stimulus; 6, no response to stimulus).
Time Frame: 6h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: The placebo group will pumped in the same volume of saline 0.9% as calculated by parturients' weight in 30 min and receive 1mg butorphanol after delivery.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Normal Saline: Drug: Normal saline control group receive NS after delivery. Drug: butorphanol tartrate PCA: butorphanol tartrate after cesarean section.
- Dexmedetomidine 0.03ug/kg/h Group: This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min and 1mg butorphanol tartrate after delivery.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.03ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Dexmedetomidine 0.03ug/kg/h: Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.03ug/kg/h Dexmedetomidine after cesarean section.
- Dexmedetomidine 0.05ug/kg/h Group: This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min and 1mg butorphanol tartrate after delivery.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.05ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Dexmedetomidine 0.05ug/kg/h: Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.05ug/kg/h Dexmedetomidine after cesarean section.
- Dexmedetomidine 0.08ug/kg/h Group: This group will receive 0.5ug/kg intravenous dexmedetomidine diluted to 4ug/ml in 30 min and 1mg butorphanol tartrate after delivery.
  Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate with 0.08ug/kg/h dexmedetomidine, diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Dexmedetomidine 0.08ug/kg/h: Drug: Dexmedetomidine This group receive Dex 0.5ug/kg after delivery. Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.08ug/kg/h Dexmedetomidine after cesarean section.
Arm/Group | Control Group | Dexmedetomidine 0.03ug/kg/h Group | Dexmedetomidine 0.05ug/kg/h Group | Dexmedetomidine 0.08ug/kg/h Group
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 2 (0) | 2.17 (0.38) | 2.14 (0.35) | 3.14 (0.71)

5. Secondary Outcome: The Degree of Satisfaction
Description: The degree of satisfaction (0, very satisfied; 1, satisfied; 2, moderately satisfied; 3, not satisfied) was evaluated at 48 h after surgery. The number of overall satisfied patients (satisfied and very satisfied) is reported.
Time Frame: 48h after cesarean section.
Measure: Count of Participants; unit: Participants
Groups:
- Group C: This group will receive 30 ml 0.9% sodium chloride in 30 min. Postoperative analgesic formula: 3ug/kg/h butorphanol tartrate diluted with normal saline to 100ml. Background dose: 2ml/h, PCA: 0.5ml, locking time: 15 min.
  Drug: butorphanol tartrate and Dexmedetomidine. PCA: butorphanol tartrate with 0.03ug/kg/h Dexmedetomidine after cesarean section.
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
Participants | 12 | 16 | 26 | 25

6. Secondary Outcome: Number of Participants That Experienced Nausea or Vomiting
Description: Total times during 48h after cesarean section.
Time Frame: 48h after cesarean section.
Measure: Number; unit: participants
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
participants | 1 | 2 | 1 | 1

7. Secondary Outcome: Ramsay Sedation Score(RSS)
Description: Sedation intensity measured with RSS is recorded at the 6, 12, 24, and 48 h after cesarean section. Sedation was assessed by the Ramsay Sedation Scores (RSS) (1, anxious patient; 2, cooperative and tranquil; 3, responding to command; 4, brisk response to stimulus; 5, sluggish response to stimulus; 6, no response to stimulus).
Time Frame: 12h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 2 (0) | 2.21 (0.41) | 2.28 (0.45) | 3.21 (0.74)

8. Secondary Outcome: Ramsay Sedation Score(RSS)
Description: as for outcome 7
Time Frame: 24h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 2 (0) | 2.07 (0.26) | 2.10 (0.31) | 2.25 (0.44)

9. Secondary Outcome: Ramsay Sedation Score(RSS)
Description: as for outcome 7
Time Frame: 48h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 2 (0) | 2 (0) | 2 (0) | 2 (0)

10. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) at Rest
Description: as for outcome 1
Time Frame: 24h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 3.21 (0.92) | 2.93 (1.03) | 1.72 (0.84) | 1.57 (1.17)

11. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS)
Description: as for outcome 1
Time Frame: 48h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 2.11 (0.96) | 2 (0.8) | 1.72 (0.84) | 125 (0.75)

12. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) on Movement
Description: visual analogue scale (VAS; with 0, no pain; to 10, the worst imaginable pain) is a validated assessing scale for pain intensity. VAS on movement was assessed when patients changed from supine to lateral position.
Time Frame: 6h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 4.39 (0.74) | 4.31 (1.14) | 2.86 (1.48) | 2.2 (0.65)

13. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) on Movement
Description: as for outcome 12
Time Frame: 12h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 3.71 (0.81) | 3.52 (0.87) | 2.69 (1.07) | 1.18 (0.86)

14. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) on Movement
Description: as for outcome 12
Time Frame: 24h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 3.82 (0.86) | 3.79 (0.82) | 2.35 (1.20) | 1.93 (1.02)

15. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) on Movement
Description: as for outcome 12
Time Frame: 48h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 3.43 (1.26) | 3.28 (1.10) | 2.24 (1.19) | 1.21 (0.92)

16. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) on Uterine Cramping
Description: visual analogue scale (VAS; with 0, no pain; to 10, the worst imaginable pain) is a validated assessing scale for pain intensity. VAS-C was assessed when the patient required oxytocin after surgery in supine position
Time Frame: 6h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 3.86 (0.85) | 3.66 (0.94) | 2.79 (0.98) | 2 (1.22)

17. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) on Uterine Cramping
Description: as for outcome 16
Time Frame: 12h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 3.46 (1.20) | 3.41 (0.95) | 2.17 (1.00) | 1.07 (1.15)

18. Secondary Outcome: Postoperative Pain Score (Visual Analogue Scale, VAS) on Uterine Cramping
Description: as for outcome 16
Time Frame: 24h after cesarean section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group C | Group D1 | Group D2 | Group D3
Number analyzed (Participants) | 28 | 29 | 29 | 28
score on a scale | 3.75 (1.35) | 3.55 (0.99) | 2.59 (1.21) | 1.79 (1.10)

ADVERSE EVENTS:
Time Frame: Every 6 hours post cesarean section, up to 48 hours in total.
Arm/Group | Group C | Group D1 | Group D2 | Group D3
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29 | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 1/28 | 2/29 | 1/29 | 1/28
OTHER ADVERSE EVENTS (reported when occurring in more than 4.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group C (N=28) | Group D1 (N=29) | Group D2 (N=29) | Group D3 (N=28)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT03065530/Prot_SAP_000.pdf